CLINICAL TRIAL: NCT00942474
Title: A Prospective, Non Randomized, Single-center, Non-blinded Feasibility Study Examining the Use of a Nerve Access Tool
Brief Title: Nerve Access Tool Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Medtronic made a business decision to discontinue the study and withdraw the IDE.
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: #1632
Record Dates: First submitted 2009-07-20; First posted 2009-07-21 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Cystocele
Keywords: The focus of the study is to assess the ability of the nerve access tool to facilitate nerve lead placement
MeSH Terms: conditions — Cystocele

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Research Arm (Experimental): Facilitate nerve stimulation lead placement with the nerve access tool
  Interventions: Device: Facilitate nerve stimulation lead placement with the nerve access tool

INTERVENTIONS:
Device: Facilitate nerve stimulation lead placement with the nerve access tool

SUMMARY:
The purpose of this study is to assess the ability of the nerve access tool to facilitate nerve stimulation lead placement.

ELIGIBILITY:
Inclusion Criteria:

* Subject is equal to or greater than 18 years of age
* Subject has a diagnosis of cystocele with planned surgical repair
* Subject has no known deficit of the nerve
* Subject is willing and able to provide written informed consent and HIPAA authorization to participate by signing the Informed Consent/Health Insurance Portability and Accountability Act Form after a full explanation of the nature and purpose of this study
* Subject is willing and able to comply with the study protocol

Exclusion Criteria:

* Subject has known neurological abnormalities of the nerve
* Subject has a known allergy to the tool or neurostimulation lead components
* Subject is pregnant or lactating

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Electromyography Response | Implant